CLINICAL TRIAL: NCT01886170
Title: Using Patient Feedback to Improve the Ways we Communicate Information Regarding Glycemic Control to Patients With Poorly Controlled Diabetes
Brief Title: Using Patient Feedback to Improve Communication Regarding Glycemic Control to Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anjali Gopalan, Robert Wood Johnson Clinical Scholar, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 817693; 00000notapplicable (Other Grant/Funding Number: UPenn Dept of Medical Ethics and Health Policy)
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes
Keywords: Adults with self-reported diagnosis of diabetes recruited from waiting rooms at outpatient primary care sites at the University of Pennsylvania
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hemoglobin A1C (No Intervention): The arms apply to the second phase of the study. This is the control arm. Participants will receive information regarding their diabetes control using the hemoglobin A1C value (standard medical information)
- Experimental Format #1 (Experimental): In phase II of the study, participants in this arm will receive information about their current diabetes control conveyed using experimental format #1. The experimental formats will be determined based on the results from Phase I of the study.
  Interventions: Other: Phase II of the Study: Information regarding Current Diabetes Control
- Experimental Format #2 (Experimental): In phase II of the study, participants in this arm will receive information about their current diabetes control conveyed using experimental format #2. The experimental formats will be determined based on the results from Phase I of the study.
  Interventions: Other: Phase II of the Study: Information regarding Current Diabetes Control

INTERVENTIONS:
Other: Phase II of the Study: Information regarding Current Diabetes Control — Participants will receive information regarding their current diabetes control in different ways depending on their assigned study arm.
  Arms: Experimental Format #1; Experimental Format #2

SUMMARY:
In this two-phase mixed methods study, the investigators will first use patient feedback from semi-structured interviews to explore the ways in which patients with diabetes understand their diabetes and assess their disease control. The investigators will also use these interviews to elicit patient feedback on promising alternative communication formats to the hemoglobin A1C (A1C). In the second phase of the study, the investigators will test new formats to communicate information regarding diabetes control to patients with poorly controlled diabetes. This phase will be a three arm RCT comparing the effect of A1C (standard medical information) versus two alternative formats on several participant outcomes, primarily glycemic control at 6 months post-intervention.

DETAILED DESCRIPTION:
The noted importance of understanding glycemic control is concerning given studies estimating that only 25% of patients understand the hemoglobin A1C value (A1C). The A1C is a blood test value reflecting average blood sugars over the previous 3 months and is used as both a clinical indicator of diabetes control with guideline-set targets and as a communication format to express level of disease control to patients.Past work has demonstrated the potential effectiveness of translating poorly understood medical values, like the A1C, into more universally understood forms. We believe applications can be used to address the problem of the poorly understood A1C. This study is two-phase mixed methods approach. We will design alternative communication formats to convey the information provided by the A1C to patients and evaluate the effectiveness of these formats in improving glycemic control, increasing patient understanding of their diabetes control, and altering patient behaviors. In Phase I of the study,we will use patient feedback from semi-structured interviews with 17-25 patients with diabetes to explore the ways in which patients assess and gauge their diabetes control, as well as to elicit patient feedback on promising communication formats. Potential alternative communication formats include categories represented by color-based scales (red/yellow/green), comparisons to averages or norms, trajectories of control over time and modified medical terminology (i.e., changing the name of the test). In phase II, patients with poorly controlled diabetes will be randomized to receive information on their glycemic control through one of three study arms, A1C (control) or one of two experimental format arms (chosen based on phase I results) and the effects of these different communication formats will be evaluated.

ELIGIBILITY:
For Phase I:

Inclusion Criteria:

* Adults who report a diagnosis of diabetes

Exclusion Criteria:

* People without diabetes

For Phase II:

Inclusion Criteria

-Adults seen at University of Pennsylvania primary care practice with a diagnosis of diabetes documented in the electronic health record and a recent hemoglobin A1C >8 %

Exclusion

* No diabetes
* No A1C or recent A1C <8%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
For Phase I of the Study: Metrics Used to Understand Diabetes Control | 4 months
  Identification of common factors patients use to understand their diabetes and diabetes control via a qualitative analysis of the patient interview responses
For Phase II of the Study: Change in Hemoglobin A1C | 6 months following enrollment
  Change in A1C between enrollment and 6-months compared between study arms.

SECONDARY OUTCOMES:
For Phase I of the study: Feedback on alternative formats | 4 months
  qualitative and quantitative analysis of the feedback received on the alternative communication formats reviewed with participants during the interviews.
For Phase II of the Study: Understanding of diabetes control | At the time of enrollment
  Accuracy of participant knowledge of level of current diabetes control

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gopalan A, Suttner L, Troxel AB, McDonough K, Schapira MM. Testing patient-informed approaches for visually depicting the hemoglobin A1c value to patients with poorly controlled diabetes: a randomized, controlled trial. BMC Health Serv Res. 2020 Mar 6;20(1):178. doi: 10.1186/s12913-020-5035-8. PMID 32143649